CLINICAL TRIAL: NCT01956968
Title: Flexibility, Range of Motion and Strength Among Patients With Differing Response to the Scapular and Humeral Assistance Tests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC13028-13KCTIL
Record Dates: First submitted 2013-09-15; First posted 2013-10-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain, Scapular dyskinesia, Physical examination
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Shoulder pain may result from abnormal arm or shoulder blade (scapular) movement. These abnormal movements may result from a variety of flexibilty, motion or strength impairments. Therefore identifying any abnormal arm or scapular movement, as well as any impairments that are associated with them can help clinicians plan a proper management strategy for patients presenting with shoulder disorders. Our hypothesis is that specific impairments will be associated with abnormal arm movement, while other impairments will be associated with abnormal scapular movement among patients with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, main complaint of shoulder pain, ability to elevate arm in the scapular plane to at least 135 degrees, pain during scapular plane elevation, can read Hebrew.

Exclusion Criteria:

* Signs or symptoms suggesting cervical spine origin, previous fracture around shoulder complex, traumatic onset of shoulder pain, Fibromyalgia, Rheumatiod arthritis, previous shoulder surgery, loss of 50% or more of passive range of motion in 2 or more planes of motion, positive lag signs, positive apprehension test, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 subjects referred to physical therapy due to shoulder pain.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | Baseline
  Measurement of supine glenohumeral internal rotation range of motion.
Posterior capsule flexibility | Baseline
  Measurement of sidelying glenohumeral horizontal adduction
Pectoralis minor resting length | Baseline
  Distance from coracoid process to 4th rib attachment onto sternum
Scapular dyskinesis | Baseline
  Visual assessment and classification of scapular movement pattern
Scapular upward rotation range of motion | Baseline
  Measured by the use of an inclinometer placed on top of scapular spine during various degrees of glenohumeral elevation angles.
Shoulder elevation torque | Baseline
  Measured with a hand-held dynamometer
Shoulder external rotator torque | Baseline
  Measured with a hand-held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Alon Rabin, PhD, Study Director — Ariel University
Locations (1):
- Bat-Yamon Physical Therapy Clinic - Clalit Health Services, Bat Yam, Israel